CLINICAL TRIAL: NCT05479968
Title: Spectroscopic Assessment of Intramyocardial Oxygen Saturation Feasibility During Open-heart Surgery
Status: Completed | Type: Observational
Sponsor: Spectrocor (Industry)
Collaborators: Hospital District of Helsinki and Uusimaa (Other)
Responsible Party: Sponsor
Other Study IDs: Safe-op 1.0
Record Dates: First submitted 2021-09-07; First posted 2022-07-29 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Coronary Artery Disease; Heart Valve Diseases
Keywords: Monitoring, Intraoperative; Heart Surgery
MeSH Terms: conditions — Coronary Artery Disease; Heart Valve Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Tissue Spectrometry group: The experimental group is subjected to testing the Specrocor Investigational Device.
  Interventions: Device: Spectrocor device

INTERVENTIONS:
Device: Spectrocor device — This feasibility study is intended to document the feasibility, safety, and usability of the Investigational device.

SUMMARY:
This traditional feasibility study aims to capture preliminary safety and effectiveness information on a near-final Investigational Device design to adequately plan the forthcoming pivotal study.

DETAILED DESCRIPTION:
The study design is based on measuring the depth of ischemia during the operation, which is compared to the intraoperative and postoperative morbidity of the patient, especially to the dysfunction of the heart.

A qualified and experienced Monitor is assigned for the study to oversee and document the progress of the trial. The Monitor ensures the trial performance in accordance with the Protocol and Good Clinical Practice (GCP).

The trial team conforms to ISO 13485 quality standards and ISO 14155 GCP. Processes included in the monitoring activities are documented in the quality management system. Below are described the summaries of all these activities.

Source data will be collected and transferred into the electronic CRFs by site staff, and the collected data quality and the conformity to the Good Clinical Practice will be assessed by monitoring. Based on a risk assessment performed, a Data Monitoring Committee shall not be established.

Clinical Research Associate (CRA) is responsible for checking the accuracy and completeness of Case Report Form (CRF) entries, source documents, and other investigation-related records against each other. Other responsibilities of CRA, including detailed Source Data Verification (SDV), are documented by the clinical project manager (CPM) or head of clinical research (HCR)(both are sponsor's representatives). SDVs will be performed and documented during monitoring visits.

Monitoring planning, reporting, and visits are pre-defined and documented with pre-made templates per the sponsor's quality management system. Monitoring visits will be performed to cover data from all study participants, and according to QMS and the Standard Operation Procedures.

The monitoring shall ensure that all source documentation is precise and document control is exercised in all relevant documentation. The monitoring ensures, that the Adverse events are always reported and appropriate authorities or stakeholders are informed.

ELIGIBILITY:
Inclusion Criteria:

* Any 18 to 90-year old patient scheduled for open-heart operation
* The ability to understand the objective of the study and the risks involved.
* Informed consent obtained, including the agreement to authorization to use the protected personal patient records according to privacy legislation.

Exclusion Criteria:

* Inability to obtain an informed consent form
* Patients included as vulnerable population according to Finnish Medical Research Act, including retarded, pregnant women, nursing mothers, prisoners, or forensic patients.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for open-heart operation
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2021-09-10 (Actual); Primary Completion 2022-01-24 (Actual); Study Completion 2022-01-24 (Actual)

PRIMARY OUTCOMES:
Number of participants with device-related adverse events as assessed by CTCAE v4.0 | Day 1-14 During hospitalization
  This traditional feasibility study aims to capture preliminary safety and effectiveness information on a near-final device design

CONTACTS AND LOCATIONS:
Overall Officials: Peter Raivio, Principal Investigator — Section Chief of Department, Head and Lung Center, Hospital District of Helsinki and Uusimaa
Locations (1):
- Heart and Lung Center, Helsinki, Uusimaa, Finland

IPD SHARING:
Plan to Share IPD: No